CLINICAL TRIAL: NCT03295331
Title: A Non-Interventional Retrospective Study To Assess The Level Of Asthma Control Among Adults at 2 Tertiary Care Centres In Malaysia
Brief Title: Assessment of Asthma Control Level in Malaysia
Acronym: ASCORE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00116
Record Dates: First submitted 2017-08-29; First posted 2017-09-27 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Asthma Control Level

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GINA-defined clinical diagnosis of Asthma: All patients with GINA-defined clinical diagnosis of Asthma seen at respiratory clinic from January to August 2016 with age 18 and above

SUMMARY:
A Non-Interventional Retrospective Study To Assess The Level Of Asthma Control Among Adults at 2 Tertiary Care Centres In Malaysia; Institute Of Respiratory Medicine (IPR) And Hospital Serdang. The specific objective of the study is to assess, in real-life clinical practice in Malaysia, the level of GINA-defined asthma control and the potential risk factors for uncontrolled disease in asthma patients

DETAILED DESCRIPTION:
Despite the availability of GINA global guideline on asthma management which is widely referred by health care providers in Malaysia, the control of asthma is still a critical challenge. According to National Health and Morbidity Survey 2011, the prevalence of asthma in Malaysia is at 6.3%. Based on self-rated health status, 5.5% of patients were reported to be in good health whereas 9.9% reported poor health status although medications such as inhaled corticosteroids (ICS) and long-acting beta agonists (LABA) are widely available for effective asthma management. There is limited data to assess the level of asthma control in Malaysia which includes current clinical manifestation and future risk of exacerbation. Given the lack of data on Asthma control level, the awareness on the current disease control level will assist to properly characterise the patients based on GINA control level thus leading to appropriate diagnosis and treatment. The specific objective of the study is to assess, in real-life clinical practice in Malaysia, the level of GINA-defined asthma control and the potential risk factors for uncontrolled disease in asthma patients

ELIGIBILITY:
Inclusion Criteria:

* All patients with GINA-defined clinical diagnosis of Asthma seen at respiratory clinic from January to August 2016.
* Be at least 18 years of age

Exclusion Criteria:

* Clinical features suggesting emphysema or chronic bronchitis
* Other de-compensated organ failures

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tertiary Care Centre ( patients seen at outpatient physicians )
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Level of GINA-defined asthma control | up to 8 months
  To assess, in real-life clinical practice in Malaysia, the level of GINA-defined asthma control and the potential risk factors for uncontrolled disease in asthma patients

SECONDARY OUTCOMES:
Types of medication prescribed for asthma control | up to 8 months
  Pharmacological management used for asthma control
Asthma control level | up to 8 months
  Asthma control level measured by Asthma Control Test (ACT) score

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Institut Perubatan Respiratori, Kuala Lumpur, Kuala Lumpur
  - Hospital Serdang, Kajang, Selangor

IPD SHARING:
Plan to Share IPD: No
N/A, Non interventional Study , observational study. No patient involved

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4574&filename=ASCORE_Abstract.pdf